CLINICAL TRIAL: NCT00563472
Title: A Feasibility Study Into the Contraceptive Effect of Estetrol Alone or Combined With Either Progesterone or Desogestrel by Daily Oral Administration to Healthy Female Volunteers for 28 Days.
Brief Title: Feasibility Study Into the Contraceptive Effect of Estetrol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pantarhei Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR3081
Record Dates: First submitted 2007-11-22; First posted 2007-11-26 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: Healthy female volunteers will participate in this study
MeSH Terms: interventions — Estetrol; Desogestrel; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): 10 mg estetrol
  Interventions: Drug: estetrol
- 2 (Active Comparator): 20 mg estetrol
  Interventions: Drug: estetrol
- 3 (Active Comparator): 20 mg estetrol and 150 microg desogestrel
  Interventions: Drug: estetrol and desogestrel
- 4 (Active Comparator): 20 mg E4 and 200 mg progesterone
  Interventions: Drug: estetrol and progesterone

INTERVENTIONS:
Drug: estetrol — 10 mg orally per day for 28 days
  Arms: 1
Drug: estetrol — 20 mg orally per day for 28 days
  Arms: 2
Drug: estetrol and desogestrel — 20 mg estetrol and 150 microg desogestrel orally per day for 28 days
  Arms: 3
Drug: estetrol and progesterone — 20 mg estetrol and 200 mg progesterone orally per day for 28 days
  Arms: 4

SUMMARY:
This is an open study in 50 young, healthy, female volunteers. Women who want to participate and who are using hormonal contraception stop using their hormonal contraceptive and wait for their first spontaneous menstruation (i.e. after a wash-out cycle). Women who do not use hormonal contraception wait for their next menstruation. From the 9th day after start of the menstruation onwards follicle growth will be monitored by ultrasonography until ovulation occurs or until day 24 after start of their menses. Women who ovulate within 24 days after start of their menses will be eligible to participate and will be stratified in one of 4 groups: 10 mg estetrol (E4) alone, 20 mg E4 alone, 20 mg E4 combined with 150 mcg desogestrel and 20 mg E4 combined with 200 mg progesterone. The subjects will be treated for 28 days. Treatment will start on the first day of their menses after the pre-treatment cycle.

During the study period (28 days) the activity of the hypothalamic-pituitary-ovarian (HPO) axis will be investigated by measuring follicular development using ultrasonography and by determining serum concentrations of Follicle Stimulating Hormone (FSH), Luteinising Hormone (LH), estradiol (E2) and Progesterone (P).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years and not older than 40 years of age
* Willing to use a barrier method of contraception during the wash-out cycle, the pre-treatment cycle, the period of study drug administration, the period of lynestrenol intake (if applicable), and 14 days thereafter or until the follow-up visit if this 14-days period ends before the follow-up visit.
* Women who ovulate in the pre-treatment cycle before or on day 24 (±1) after start of their menses, who have a subsequent P concentration of > 16 nmol/l and whose next menstruation does not start within 6 days after ovulation
* Body Mass Index > 18 and <30 kg/m2
* Good physical and mental health
* Both ovaries visible upon ultrasonography
* Willing to give informed consent in writing

Exclusion Criteria:

* Clinically significant abnormal results of routine hematology, serum biochemistry, urinanalysis, and/or ECG in the opinion of the Investigator at screening.
* Known or suspected pregnancy
* Lactation
* Pregnancy during accurate hormonal contraceptive use
* Known or suspected breast cancer or a history of breast cancer
* Clinically significant abnormalities of the uterus and/or ovaries detected by examination and/or ultrasound (non-physiological ovarian mass or significant uterine pathology).
* A cervical smear with clinically relevant abnormal cytology within one year before study start.
* Previous use of depot progestogen preparations in the last 6 months.
* Contraindications for contraceptive steroids:

  * a history of, or existing thromboembolic, cardiovascular or cerebrovascular disorder
  * a history of, or existing conditions predisposing to, or being prodromi of, a thrombosis
  * a known defect in the blood coagulation system (e.g. deficiencies in AT-III, protein C, S, and APC resistance)
  * heterozygous for a mutation in coagulation factor II and/or positive for factor V Leiden
  * the presence of a severe or more than one risk factor for vascular disease (e.g. dyslipoproteinaemia; diabetes mellitus; hyperhomocysteinaemia; systemic lupus erythematosus; chronic inflammatory bowel disease; antiphospholipid antibodies; smoking; venous thromboembolism in sibling or parent below the age of 50, or arterial disease in sibling or parent below the age of 35; within 2 weeks after full remobilisation following surgery)
  * hypertension, i.e. systolic blood pressure >140 mmHg and/or diastolic blood pressure >90 mmHg
  * disturbance of liver function: e.g. cholestatic jaundice, a history of jaundice of pregnancy or jaundice due to previous oestrogen use, Rotor syndrome and Dubin-Johnson syndrome
  * known or suspected hormone-dependent tumours or endometrial hyperplasia
  * undiagnosed vaginal bleeding
  * porphyria
  * a history during pregnancy or previous hormone-use of severe pruritus, herpes gestationis or deterioration of otosclerosis
* Use of one or more of the following medications:

  * sex steroids other than the medication of study
  * use at present or within 2 months before start study medication:
  * hydantoins, barbiturates, primidone, carbamazepine, oxcarbazepine, topiramate, troglitazone, felbamate, rifampicin, rifabutin, griseofulvin and St. John's wort (Hypericum perforatum)
* Status post-partum or post-abortion within a period of 2 months before study start
* Administration of investigational drugs within 3 months before start study medication
* A history of (within 12 months) alcohol or drug abuse
* A known hypersensitivity for one of the components of the study medication (eg arachisoil and lactosis)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2007-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
ovulation inhibition | during treatment

SECONDARY OUTCOMES:
endocrine parameters | during treatment

CONTACTS AND LOCATIONS:
Overall Officials: H. Coelingh Bennink, MD, PhD, Study Director — Pantarhei Bioscience
Locations (1):
- Dinox, Groningen, Netherlands